CLINICAL TRIAL: NCT01493570
Title: Randomised, Double-blind, Placebo-controlled Parallel-group Proof of Mechanism Study to Assess the Pharmacokinetics and to Evaluate the Pharmacodynamic Effect of Different Single Oral Doses of BI 409306 in Healthy Male Volunteers
Brief Title: Assessment of Exposure of BI 409306 in Cerebrospinal Fluid (CSF) Relative to Plasma as Well as to Evaluation of the Effect of Different Doses of BI 409306 on the cGMP (Cyclic Guanosine Monophosphate) Levels in CSF in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1289.3; 2011-003749-16 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-12-12; First posted 2011-12-16 (Estimated); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — BI 409306

ARMS (5):
- BI 409306 25mg (Experimental)
  Interventions: Drug: BI 409306
- BI 409306 50 mg (Experimental)
  Interventions: Drug: BI 409306
- BI 409306 100 mg (Experimental)
  Interventions: Drug: BI 409306
- BI 409306 200 mg (Experimental)
  Interventions: Drug: BI 409306
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 409306 — Film-coated tablet
  Arms: BI 409306 100 mg; BI 409306 200 mg; BI 409306 25mg; BI 409306 50 mg
Drug: Placebo — Film-coated tablet
  Arms: Placebo

SUMMARY:
Due to the exploratory nature of this trial, there is no primary objective in a confirmatory sense. The study aims

- to evaluate the effect of different doses of BI 409306 on biomarker and to assess the exposure of BI 409306

ELIGIBILITY:
Inclusion criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs after 10 minutes in supine position (blood pressure (BP), pulse rate (PR)), body temperature (BT)), 12-lead electrocardiogram (ECG)), clinical laboratory tests
2. Age =21 and Age =50 years
3. Body Mass Index (BMI) =18.5 and BMI =29.9 kg/m2
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion criteria:

1. Any finding of the medical examination (including BP, PR and ECG) deviating from normal and considered by the investigator as clinical relevant
2. Abnormal values for Prothrombin Time (PT), (Activated Partial Thromboplastin Time (aPTT) and thrombocytes considered by the investigator as clinically relevant
3. Any evidence of a clinically relevant concomitant disease
4. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
5. Surgery of the gastrointestinal tract (except appendectomy)
6. Diseases of the central nervous system (included but not limited to any kind of seizures, stroke or psychiatric disorders)
7. History of relevant orthostatic hypotension, fainting spells or blackouts.
8. Chronic or relevant acute infections
9. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
10. Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration
11. Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
12. Participation in another trial with an investigational drug within two months prior to administration or during the trial
13. Smoker, who consume more than 5 cigarettes per day
14. Inability to refrain from smoking on trial days
15. Alcohol abuse (more than 20 g/day): 2 units/day (14 units/week)
16. Drug abuse
17. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
18. Excessive physical activities (within one week prior to administration or during the trial)
19. Any laboratory value outside the reference range that is of clinical relevance
20. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTcF interval >450 ms)
21. Inability to understand and to comply with protocol requirements and restrictions and dietary regimen of trial site
22. of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
23. Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until three month after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female (intra-uterine device with spermicide, hormonal contraceptive since at least two months)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2012-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1289.3.1 Boehringer Ingelheim Investigational Site, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomised, parallel-group, double-blinded, double-dummy, single dose trial was placebo-controlled. Test product and placebo were given as a single dose to healthy male subjects in a single centre.
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- BI 409306 25mg: Subjects were orally administered single dose of BI 409306 25 milligram (mg) (5x5 mg) film-coated tablets in the morning.
- BI 409306 50 mg: Subjects were orally administered single dose of BI 409306 50 mg (1x50 mg) film-coated tablet in the morning.
- BI 409306 100 mg: Subjects were orally administered single dose of BI 409306 100 mg (2x50 mg) film-coated tablets in the morning.
- BI 409306 200 mg: Subjects were orally administered single dose of BI 409306 200 mg (1x150 mg and 1x50 mg) film-coated tablets in the morning.
- Placebo: Subjects were orally administered BI 409306 matching placebo film-coated tablet in the morning
Period: Overall Study
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo
Started | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This analysis set included all treated subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Treated set
  Years | 39.5 (7.9) | 46.3 (2.9) | 38.5 (11.5) | 35.8 (9.0) | 29.5 (8.9) | 37.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Treated Set
  Participants
    Female | 0 | 0 | 0 | 0 | 0 | 0
    Male | 4 | 4 | 4 | 4 | 4 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Treated set
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    White | 4 | 4 | 4 | 4 | 4 | 20
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Cmax of BI 409306 in CSF Compared to Plasma
Description: Ratio of Cmax (maximum measured concentration) of BI 409306 in Cerebrospinal fluid (CSF) compared to plasma is presented. Ratio was calculated as: Cmax of BI 409306 in CSF/ Cmax of BI 409306 in plasma.
  Time frame: Blood: Within 2:00 hours (h):minutes (min) before dosing and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing.
  CSF: Within 2:00 hours (h):minutes (min) before dosing and 0:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing.
Time Frame: Pharmacokinetic samples were collected within 2 hours before and up to up to 24 hours after BI 409306 administration (please refer the description for the time frame in detail).
Population: Pharmacokinetic Set (PKS): This analysis set included all treated subjects who provided at least 1 evaluable observation for a pharmacokinetic endpoint and who had no important protocol violation relevant to the evaluation of pharmacokinetic parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
Ratio | 0.267 (18.40) | 0.244 (15.80) | 0.294 (42.80) | 0.335 (5.74)
Statistical Analysis 1: Comparison: BI 409306 25mg vs BI 409306 50 mg vs BI 409306 100 mg vs BI 409306 200 mg; Dose-adjusted CSF to plasma ratio for Cmax. The Analysis of Variance (ANOVA) model was used with 'subject nested within treatment' considered as random effect; Test type: Other; p = 1.0000, ANOVA — p-value for ratio outside interval 80% - 125%; Ratio CSF to Plasma in % = 28.31, 90% CI 2-sided [25.418 to 31.532] — Intra Individual geometric coefficient of variation (gCV [%]) = 17.50

2. Primary Outcome: Maximum Change From Baseline of cGMP in CSF Calculated as Ratio (Emax)
Description: The maximum change from baseline of cyclic guanosine monophosphate (cGMP) in cerebrospinal fluid (CSF) was calculated as: exp(ln(cGMPmax) - ln(cGMP0)), where cGMP0 is the baseline cGMP value per subject (mean of the two pre-dose measurements) and cGMPmax is the maximal cGMP value per subject measured after drug intake.
Time Frame: Within 2:00 hours (h):minutes (min) before dosing and 0:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing.
Population: Pharmacodynamic set (PDS): This analysis set included all treated subjects who provided at least 1 evaluable observation for a pharmacodynamic endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
ratio | NA (NA) — Geometric Mean (gMean) is actually adjusted gMean. GMean was adjusted for baseline cGMP concentration. Adjusted gMean = 1.826. Geometric Coefficient of Variation (gCV) is actually adjusted gCV. GCV was adjusted for baseline cGMP concentration. Adjusted gCV= 32.061 | NA (NA) — Geometric Mean (gMean) is actually adjusted gMean. GMean was adjusted for baseline cGMP concentration. Adjusted gMean = 2.254 Geometric Coefficient of Variation (gCV) is actually adjusted gCV. GCV was adjusted for baseline cGMP concentration. Adjusted gCV= 32.176 | NA (NA) — Geometric Mean (gMean) is actually adjusted gMean. GMean was adjusted for baseline cGMP concentration. Adjusted gMean = 3.030 Geometric Coefficient of Variation (gCV) is actually adjusted gCV. GCV was adjusted for baseline cGMP concentration. Adjusted gCV= 32.024 | NA (NA) — Geometric Mean (gMean) is actually adjusted gMean. GMean was adjusted for baseline cGMP concentration. Adjusted gMean = 4.864 Geometric Coefficient of Variation (gCV) is actually adjusted gCV. GCV was adjusted for baseline cGMP concentration. Adjusted gCV= 33.200 | NA (NA) — Geometric Mean (gMean) is actually adjusted gMean. GMean was adjusted for baseline cGMP concentration. Adjusted gMean = 1.478 Geometric Coefficient of Variation (gCV) is actually adjusted gCV. GCV was adjusted for baseline cGMP concentration. Adjusted gCV= 33.179

3. Primary Outcome: Maximum Relative Change From Baseline of cGMP in CSF
Description: Maximum relative change from baseline of cyclic guanosine monophosphate (cGMP) in cerebrospinal fluid (CSF) is presented.
  Maximum relative change from baseline was calculated as: (cGMPmax - cGMP0)/ cGMP0, where cGMPmax is the maximum measured concentration of cGMP after dosing of BI 409306 and cGMP0 is cGMP concentration at baseline.
Time Frame: Within 2:00 hours (h):minutes(min) before dosing and 0:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00h, 4:00, 6:00, 8:00h, 10:00, 12:00, 14:00 and 24:00 h:min after dosing.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
Ratio | 1.166 (0.714) | 1.329 (0.716) | 2.247 (0.713) | 4.973 (0.738) | 0.910 (0.737)

4. Primary Outcome: Maximum (Absolute) Change From Baseline of cGMP Concentration in CSF
Description: Maximum (absolute) change from baseline of cyclic guanosine monophosphate (cGMP) concentration in cerebrospinal fluid (CSF) is presented.
  The maximum (absolute) change from baseline in cGMP concentration was calculated as: maximum measured concentration of cGMP after dosing of BI 409306 (cGMPmax) - cGMP concentration at baseline (cGMP0).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nanomole/Liter
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
nanomole/Liter | 2.299 (0.825) | 3.451 (0.827) | 5.239 (0.824) | 9.089 (0.852) | 0.748 (0.852)

5. Secondary Outcome: Maximum Measured Concentration of BI 409306 in Plasma and CSF (Cmax)
Description: Maximum measured concentration of BI 409306 in plasma and CSF (cerebrospinal fluid) (Cmax) is reported.
  Time frame: Blood: Within 2:00 hours (h): minutes (min) before dosing and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing CSF: Within 2:00 hours (h):minutes (min before dosing and 0:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
nanomole/Liter (nmol/L)
  CSF | 46.9 (84.3) | 183 (51.3) | 271 (39.7) | 902 (36.3)
  Plasma | 176 (92.6) | 751 (35.7) | 922 (36.5) | 2700 (38.9)

6. Secondary Outcome: Time From Dosing to Maximum Measured BI 409306 Concentration in Plasma and CSF (Tmax)
Description: Time from dosing to maximum measured BI 409306 concentration in plasma and CSF (cerebrospinal fluid) (tmax) is reported.
  Time frame: Blood: Within 2:00 hours (h):minutes (min) before dosing and 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, and 24:00 h:min after dosing.
  CSF: Within 2:00 hours (h):minutes (min) before dosing and 0:00, 0:10 , 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg
Number analyzed (Participants) | 4 | 4 | 4 | 4
hour
  CSF | 2.00 [2.00 to 3.00] | 2.00 [1.00 to 2.00] | 1.75 [1.50 to 3.00] | 1.50 [0.767 to 2.02]
  Plasma | 1.25 [0.750 to 1.500] | 0.750 [0.500 to 0.750] | 0.875 [0.750 to 1.500] | 0.750 [0.483 to 1.000]

7. Secondary Outcome: Maximum Measured cGMP Concentration in CSF (Cmax)
Description: Maximum measured cyclic guanosine monophosphate (cGMP) concentration in cerebrospinal fluid (CSF) (Cmax) is reported.
Time Frame: Within 2:00 hours (h): minutes (min) before dosing and 0:00, 0:10, 0:20, 0:30, 0:45, 1:00, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00 and 24:00 h:min after dosing.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
nanomole/Liter (nmol/L) | 5.96 (3.31) | 6.32 (2.91) | 8.80 (3.44) | 11.2 (3.09) | 5.36 (1.11)

8. Secondary Outcome: Time From Dosing to Maximum Measured cGMP Concentration in CSF (Tmax)
Description: Time from dosing to maximum measured cyclic guanosine monophosphate (cGMP) concentration in cerebrospinal fluid (CSF) (tmax) is reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | BI 409306 25mg | BI 409306 50 mg | BI 409306 100 mg | BI 409306 200 mg | Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
hour | 5.00 [0.50 to 10.0] | 2.50 [1.65 to 3.00] | 3.52 [3.00 to 4.00] | 2.00 [2.00 to 4.00] | 16.00 [0.50 to 24.00]

ADVERSE EVENTS:
Time Frame: From first drug administration until end of the trial, ie., up to 17 days
Description: Treated set (TS): TS included all subjects who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Groups:
- BI 409306 50mg: Subjects were orally administered single dose of BI 409306 50 mg (1x50 mg) film-coated tablet in the morning.
- BI 409306 100mg: Subjects were orally administered single dose of BI 409306 100 mg (2x50 mg) film-coated tablets in the morning.
- BI 409306 200mg: Subjects were orally administered single dose of BI 409306 200 mg (1x150 mg and 1x50 mg) film-coated tablets in the morning.
Arm/Group | Placebo | BI 409306 25mg | BI 409306 50mg | BI 409306 100mg | BI 409306 200mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 4/4 | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | BI 409306 25mg (N=4) | BI 409306 50mg (N=4) | BI 409306 100mg (N=4) | BI 409306 200mg (N=4)
Chromatopsia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Sensation of pressure (General disorders) | 1 | 1 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 1 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 3 | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.